CLINICAL TRIAL: NCT02031263
Title: Efficacy of Bronchial Thermoplasty in Korean Patients With Severe Asthma
Brief Title: Efficacy of Bronchial Thermoplasty in Korean
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, Department of Pulmonary and Critical Care Medicine and Clinical Research Center for Chronic Obstructive Airway Diseases, Asan Medical Center, University of Ulsan College of Medicine, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thermoplasty-Br
Record Dates: First submitted 2014-01-03; First posted 2014-01-09 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- thermoplasty group (Experimental): Check on the quality of life, emergency room uses, and sudden progress of the disease of the patients before and after the treatment by using bronchial thermoplasty system by using paired t test.
  Interventions: Procedure: bronchial thermoplasty system

INTERVENTIONS:
Procedure: bronchial thermoplasty system — Check on the quality of life, emergency room uses, and sudden progress of the disease of the patients before and after the treatment by using bronchial thermoplasty system by using paired t test.
  Other Names: ALAIR

SUMMARY:
The investigators will find out if bronchial thermoplasty shows efficacy in reducing acute exacerbation and improving quality of life for uncontrolled asthma in Korea through this research. US FDA approved this procedure and CE mark was taken in Europe. Many procedure was performed in Western countries.

Korean FDA have approved this procedure in 2013. However, no procedure was performed in Korea, and the data is rare in Asian countries. In this study, investigators will examine the efficacy of this procedure in Korean asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* 1) Eighteen-year-old or older
* 2) Patients whose asthma is not controlled with more than three months of using high dose inhaled steroids and long acting β2-agonists
* 3) Patients with pre-bronchodilator FEV1 is between sixty and eighty-five%
* 4) Patients who do not improve through continuous drug uses.

Exclusion Criteria:

* 1) Presence of a pacemaker, internal defibrillator, or other implantable electronic devices,
* 2) Known sensitivity to medications required to perform bronchoscopy, including lidocaine, atropine, and benzodiazepines.
* 3) Patients previously treated with the Alair System should not be retreated in the same area(s). No clinical data are available studying the safety and/or effectiveness of repeat treatments.
* 4)Active respiratory infection
* 5) Asthma exacerbation or changing dose of systemic corticosteroids for asthma (up or down) in the past 14 days.
* 6) Known coagulopathy.
* 7) As with other bronchoscopic procedures, patients should stop taking anticoagulants, antiplatelet agents, aspirin and NSAIDS before the procedure with physician guidance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Questionnaire for Adult Korean Ashtmatics - QLQAKA Questionnaire for Adult Korean Ashtmatics - QLQAKA | 3 months

SECONDARY OUTCOMES:
Quality of Life Questionnaire for Adult Korean Ashtmatics - QLQAKA Questionnaire for Adult Korean Ashtmatics - QLQAKA | 6 months
Acute exacerbation | 3,and 6 months
  Acute exacerbation of asthma is defined as following: episodes of progressive increase in shortness of breath, cough, wheezing, or chest tightness, or some combination of these symptoms leading change of medications (use of systemic steroids or antibiotics)

CONTACTS AND LOCATIONS:
Overall Officials: Sei Won Lee, MD, Principal Investigator — Department of Pulmonary and Critical Care Medicine and Clinical Research Center for Chronic Obstructive Airway Diseases, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Republic of Korea
Locations (1):
- Department of Pulmonary and Critical Care Medicine and Clinical Research Center for Chronic Obstructive Airway Diseases, Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea